CLINICAL TRIAL: NCT02846012
Title: Prospective Observational Study Utilizing Next Generation Continuous Single Culture Media (CSCM2) for Comparative in Vitro Embryo Development and Outcome Data
Brief Title: Comparison of Culture Media for in Vitro Embryo Development
Acronym: NXGeM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ovation Fertility (Other)
Responsible Party: Principal Investigator, Matthew VerMilyea, Laboratory Director, Ovation Fertility
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-NxGeM-01
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSCM Control (No Intervention): Control medium
- CSCM2 (Experimental): New Formulation medium
  Interventions: Other: CSCM2

INTERVENTIONS:
Other: CSCM2
  Arms: CSCM2

SUMMARY:
The purpose of this study is to collect development and outcome data on human embryos which are cultured in a 2nd generation continuous single culture medium (CSCM2) with the objective to demonstrate its performance efficacy in comparison to existing commercially available single culture or continuous embryo culture media.

DETAILED DESCRIPTION:
A multi-center (3 sites and 2 investigators), prospective trial with up to 300 patients. Patients will be enrolled from participating sites from the United States. Study sites will conduct this study under the oversight of Sterling IRB. Each study site should enroll enough patients to achieve at least 50 evaluable patients that have undergone a treatment cycle using split case sibling embryos in which half of the embryos are cultured in CSCM2 and the other half in current CSCM (as control).

The methods will consist of standard ovarian stimulation protocols at each facility to obtain a sufficient number of mature (MII) oocytes for fertilization by ICSI. Following fertilization, identified diploid (2PN) zygotes will be evenly divided and randomly allocated to the embryo culture treatment conditions of CSCM2 or CSCM and cultured according to standard laboratory procedure (incubated in 5-6% CO2 in air or low O2 concentrations of 5-6%) to the blastocyst stage (Day 5/6 or 7). Top quality blastocyst(s) will be transferred and monitored for implantation, pregnancy and ongoing birth. Embryo transfers will either occur in a fresh or frozen cycle.

The procedures in this study are designed to follow the standard medical care at each study site for women having IVF treatment (the participant will sign a separate consent at your clinic for your IVF procedures). The participants study doctor will explain in detail the procedures participants will undergo at the clinic; this form is only meant to explain the details of the research study. This study does not involve randomization of patient participation or any sham procedures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age in good general physical and mental health.
* Women undergoing fresh in vitro fertilization treatment using their own eggs which will be fertilized by ICSI only
* Normal uterine cavity, as defined by the program.
* Normal BMI (< 35).
* Normal endocrine workup (including PCOS patients).
* Fresh or Frozen Blastocyst transfer
* At least 4 diploid zygotes showing signs of normal (2PN) fertilisation
* Willing to have half of their 2PN embryos cultured in CSCM and the other half of their 2PN embryos cultured in CSCM 2nd generation
* Willing to comply with study protocol and procedures
* Willing to provide written informed consent

Exclusion Criteria:

* Use of donor egg / gestational carrier
* Couples for whom the male partner requires surgically extracted sperm (testicular or epididymal retrieval)
* History of complications related to tolerance to OCP's, Gonadotropins, Progesterone or estrogen.
* A medical condition that is contraindicated to pregnancy or gonadotropin therapy (eg. allergies, immune deficiency, etc.)
* History of cancer

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Pregnancy Success | 2 years
  Live Birth

SECONDARY OUTCOMES:
Implantation | 2 years
  Presence of Gestational Sac
Embryo Development | 2 years
  Blastocyst Utilisation Rate (number of fertilised embryos which develop to usable blastocysts)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew VerMilyea, PhD, Principal Investigator — Ovation Fertility
Locations (1):
- Ovation Fertility - Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, however, collated data may be used for publication without patient identification.